CLINICAL TRIAL: NCT07043231
Title: Evaluation of Creative Materials Supporting Healthcare Professionals in Discussing Suicidality in Children and Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Flemish Minister for Welfare, Public Health and Family, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0593
Record Dates: First submitted 2025-05-27; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental)
  Interventions: Other: Creative materials

INTERVENTIONS:
Other: Creative materials — This intervention provides professionals with co-created creative materials specifically designed to facilitate structured, safe conversations about suicidality with children and adolescents. Unlike standard tools, it offers three flexible pathways-Conversation, Drawing, and Walking-allowing a personalized approach tailored to the young person's preferences and context. The materials guide professionals through the assessment of suicidal intent, risk and protective factors, and help formulate a risk assessment and Safety Plan. The content is aligned with national clinical guidelines but uniquely integrates experiential insights from youth with lived experience, ensuring both theoretical grounding and practical applicability.

SUMMARY:
Preliminary research clearly indicates a significant shortage of evidence-based tools and interventions specifically targeting suicidality among children and adolescents. The need for such methodologies is substantial, as suicidal ideation and suicide attempts are relatively common within this age group. According to the 2022 Health Behaviour in School-aged Children (HBSC) study, 16% of boys and 28% of girls aged 13 to 18 reported having had suicidal thoughts on two or more occasions in their lifetime (Schrijvers et al., 2023). Compared to the previous HBSC study conducted in 2018, this represents a negative trend, as 13% of boys and 22% of girls reported suicidal thoughts at that time (Dierckens et al., 2019).

Facilitating open discussions about suicidal thoughts is therefore of critical importance. Research has shown that discussing suicidality does not increase suicidal behavior; rather, it can contribute to a reduction in risk (Blades et al., 2018; Dazzi et al., 2014; DeCou & Schumann, 2018; Polihronis et al., 2022). Breaking the taboo around suicidality and attuning to the emotional experiences of children and adolescents may serve as an initial step toward providing effective support. Such openness can help reduce feelings of loneliness and isolation by fostering a safe environment in which young people feel heard and understood. Moreover, the act of speaking openly about suicidality is associated with increased social support-an important protective factor (Batty et al., 2018; Calati et al., 2019).

In 2023, a project was launched aimed at developing creative materials to support professionals in initiating conversations about suicidality with children and adolescents. This material is being developed through a co-creative process (EC code: ONZ-2024-0211), in collaboration with youth care professionals, method developers, and young individuals with lived experience of suicidal thoughts. These young people provide essential contributions to ensure that the materials are aligned with their needs and expectations for support. This co-creative approach aims not only to produce a theoretically grounded methodology, but also to yield a practically applicable tool that effectively addresses the real-world challenges faced by both professionals and youth. The creative materials are currently under development and are designed to facilitate exploration and discussion of suicidality, ultimately supporting professionals in formulating a risk assessment and developing a Safety Plan. This approach aligns with the recommendations outlined in the guideline "Detection and Interventions for Suicidal Thoughts and Behaviors in Children and Adolescents" (Dumon et al., 2023).

The next phase of the project focuses on evaluating the creative materials. The evaluation aims to gain insight into their usability and applicability in professional practice. This will be conducted through an evaluation study. Professionals working in Flanders will be recruited via calls on www.zelfmoord1813.be, relevant partner organizations, social media, and newsletters from VLESP and other partners. Additionally, professionals may be invited via email. Those who have used the materials over a three-month period will be asked to retrospectively share their experiences. The study consists of the following steps:

Registration: Eligible professionals complete a short registration form (duration: approximately 5 minutes).

Use of the creative materials: Participants use the materials in their professional context over a period of three months.

Post-assessment: At the end of the three-month period, participants complete a questionnaire regarding their experiences with the materials (duration: approximately 10-15 minutes).

The post-assessment focuses on evaluating user-friendliness, practical applicability, and the potential of the creative materials to facilitate conversations about suicidality. Collected feedback will be used to further refine and optimize the materials. If participants do not complete the post-assessment promptly, they will receive reminder emails after 2 and 4 days. The target sample size for the study is 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthcare professionals (e.g., general practitioners, psychiatrists, psychologists, psychotherapists, or nurses) working in mental health care.
* Participants must work with children or adolescents who may be experiencing suicidality.
* Participants must be 18 years of age or older.
* Participants must have internet access and sufficient proficiency in Dutch.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Usability of Creative Materials for Discussing Suicidality | Three months after enrollment
  This is self-developed questionnaire regarding the usability of the creative materials.

SECONDARY OUTCOMES:
Efficacy of Creative Materials for Discussing Suicidality | Three months after enrollment
  This is a self-developed questionnaire regarding the efficacy of the creative materials.
Applicability of the creative materials for Discussing Suicidality | Three months after enrollment
  This is a self-developed questionnaire regarding the applicability of the creative materials.
Acceptability of Intervention Measure (AIM) | Three months after enrollment
  This is a psychometrically validated tool developed by Weiner et al. (2017) which assesses the perceived acceptability of an intervention by stakeholders. The measure consists of 4 items, rated on a Likert scale (typically 1 = completely disagree to 5 = completely agree).
Intervention Appropriateness Measure (IAM) | Three months after enrollment
  This is a psychometrically validated tool developed by Weiner et al. (2017) which evaluates the perceived relevance or suitability of the intervention for a given setting or problem. The measure consists of 4 items, rated on a Likert scale (typically 1 = completely disagree to 5 = completely agree).
Feasibility of Intervention Measure (FIM) | Three months after enrollment
  This is a psychometrically validated tool developed by Weiner et al. (2017) which measures the extent to which an intervention can be successfully used or carried out within a setting. The measure consists of 4 items, rated on a Likert scale (typically 1 = completely disagree to 5 = completely agree).
Implementation of the creative materials for Discussing Suicidality | Three months after enrollment
  This is a self-developed questionnaire regarding the implementation of the creative materials.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — University Ghent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium